CLINICAL TRIAL: NCT04475965
Title: The Influence of the Intensity of Isometric Exercise on Pain Intensity, Muscle Pain Sensitivity and Function in Patients With Chronic Shoulder Pain: A Parallel Single-blind Randomized Study
Brief Title: The Effectiveness of Isometric Exercise on the Management of Chronic Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jorge Fuentes (Other)
Responsible Party: Sponsor-Investigator, Jorge Fuentes, Clinical professor, Universidad Católica del Maule
Organization: Universidad Católica del Maule (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EIH UCM
Record Dates: First submitted 2020-07-13; First posted 2020-07-17 (Actual); Last update posted 2020-07-17 (Actual); Status verified 2020-07

CONDITIONS: Chronic Shoulder Pain
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to groups by using a random number table. This procedure was conducted by an external assessor. The allocation concealment strategy included the use of sealed-opaque and consecutively numbered envelopes.
Who Masked: Outcomes Assessor
Masking Description: The assessor responsible for the outcome measures was blinded to the subjetc´s treatment assignment. The assessor was not present in the room while the treatment was delivered. He returned once the treatment was completed to perform the measurements.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 20% maximal voluntary isometric contraction (Experimental): Patients in group 1 received a five-series Isometric Contraction of shoulder external rotators at 20% of maximal voluntary isometric contraction. Each series of Isometric Contraction was done until exhaustion or up to a maximum of 5 minutes. Patients received five sessions of treatment during a two-week period.
  Interventions: Other: Isometric exercise for shoulder external rotators
- Group 2 80% maximal voluntary isometric contraction (Active Comparator): Patients in group 2 received a five-series Isometric Contraction of shoulder external rotators at 80% of maximal voluntary isometric contraction. Each series of Isometric Contraction was done until exhaustion or up to a maximum of 5 minutes. Patients received five sessions of treatment during a two-week period.
  Interventions: Other: Isometric exercise for shoulder external rotators

INTERVENTIONS:
Other: Isometric exercise for shoulder external rotators — The intervention included the application of a series of isometric contraction for the external rotators shoulder muscles. The exercise protocol included two intensities; high-level isometric contraction (80% maximal voluntary isometric contraction) versus a low-level isometric contraction (20% maximal voluntary isometric contraction).

SUMMARY:
The aim of this study was to evaluate the influence of the intensity of Isometric Contraction of shoulder external rotators, comparing the effect of a high-level IC (80% maximal voluntary isometric contraction) versus a low-level Isometric Contraction (20% maximal voluntary isometric contraction) on pain intensity, pain thresholds, and function in chronic pain shoulder patients.

DETAILED DESCRIPTION:
This was a single-blinded, randomized parallel study. Eighty-two patients presenting chronic musculoskeletal shoulder pain were allocated to two groups. Patients in group 1 (n= 41) received a five-series Isometric Contraction of shoulder external rotators at 20% maximal voluntary isometric contraction, while patients in group 2 (n= 41) received similar protocol but the intensity of contraction was set at 80% maximal voluntary isometric contraction. In both cases, each series of IC was done until exhaustion or up to a maximum of 5 minutes. Patients received five sessions of treatment during a two-week period. Outcome measures included muscle pain sensitivity (pressure pain thresholds) and pain intensity (pain intensity numerical rating score), and shoulder function (Constant Score).

ELIGIBILITY:
Inclusion Criteria:

* Male or female having a chronic shoulder soft-tissue injury of at least 3 month duration resulting in a mild to moderate level of disability (Constant score scale), pain intensity score between 3 and 8 points (pain intensity numerical rating scale), and age between 18 and 65 years.

Exclusion Criteria:

* Participants were excluded if they had any contraindications related to the application of isometric exercise, neurological problems (central or peripheral), concomitant physiotherapy or chiropractic treatment, fibromyalgia or general systemic disease conditions, had participated in any moderate or vigorous physical activity in the las 72 hours previous the outcome assessment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-08-27 (Actual); Study Completion 2019-10-05 (Actual)

PRIMARY OUTCOMES:
Pain intensity Numerical Rating Scale | Baseline through the end of the intervention (2 week period)
  The Pain intensity Numerical Rating Scale is a self-reporting measure of pain intensity. This involves asking patients to rate their pain intensity by selecting a number on a horizontally depicted 11-point scale from 0 (no pain) to 10 (worst possible pain). Based on its several advantages (i.e. more responsive, sensitive and easy to administer) over other pain measuring scales, the PI-NRS has been recommended as a core outcome measure in clinical trials of chronic pain treatments. The minimal clinically important change for this scale has been reported to range from 1.5 to 3.2 points. Other authors have determined a meaningful clinical change of 2 points from baseline pain scores.

SECONDARY OUTCOMES:
Shoulder function | Baseline through the end of the intervention (2 week period)
  The shoulder function was assessed by the Constant Score scale. This is a multi-item functional scale assessing pain, activities of daily living, range of motion and strength of the affected shoulder. Its score ranges from 0 to 100 points, representing worst and best shoulder function respectively.
  Pain and activities of daily living (subjective aspects receiving 35 points) are answered by the patient ; and range of motion and strength (objective aspects receiving 65 points) require a physical evaluation and are answered by the orthopaedic surgeon or the physiotherapist.
Muscle pain sensitivity | Baseline through the end of the intervention (2 week period)
  Muscle pain sensitivity was evaluated through the pressure pain threshold, or the minimum pressure that induces pain or discomfort. Pressure pain thresholds measurements have been shown to have good or excellent inter-rater intraclass correlation coeficient values ranging from 0.74 to 0.90, and intra-rater reliability interclass correlation coefficient values ranging from 0.75 to 0.99. The minimal clinically important change calculated for this outcome has been reported to be ≥ 1.10 Kg/cm2/s

CONTACTS AND LOCATIONS:
Overall Officials: Hans Neira, BSc, Principal Investigator — Concepcion University
Locations (1):
- Hospital Traumatológico, Concepción, Bio Bio, Chile

IPD SHARING:
Plan to Share IPD: No